CLINICAL TRIAL: NCT01381523
Title: A Combination Product of Sumatriptan and Naproxen Sodium Versus Single-entity Oral Triptans: An Analysis of Real World Data
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113913
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Migraine Disorders
Keywords: resource utilization; naproxen sodium; cost and cost analysis; triptan; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Combined Modality Therapy; Sumatriptan; Naproxen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study-treatment naive insured adults with migraine: Adult health care plan members with a pharmacy claim for a combination product of sumatriptan and naproxen sodium (SumaRT/Nap) and propensity score matched controls with a pharmacy claim for a single-entity triptan
  Interventions: Drug: Combination therapy with sumatriptan and naproxen sodium (SumaRT/Nap); Drug: Single-entity oral triptans
- Insured adults with migraine who switch study treatment: Adult health plan members with a pharmacy claim for SumaRT/Nap following at least one single-entity triptan pharmacy claim in the previous 6 months and propensity-score matched controls who switched from one single-entity triptan to another
  Interventions: Drug: Combination therapy with sumatriptan and naproxen sodium (SumaRT/Nap); Drug: Single-entity oral triptans

INTERVENTIONS:
Drug: Combination therapy with sumatriptan and naproxen sodium (SumaRT/Nap) — Patients with new pharmacy claims for SumaRT/Nap with separate analyses for patients with at least one triptan pharmacy claim in the 6-month, pre-index period and those who are triptan-naive based on 6 months of data
  Other Names: Treximet® is a registered trademark of GlaxoSmithKline
Drug: Single-entity oral triptans — Patients are propensity score matched to patients in the SumaRT/Nap groups and analyzed separately if patient has a pharmacy claim for a different type of triptan in the previous 6 months or is triptan treatment naive. Triptans included almotriptan, naratriptan, rizatriptan, eletriptan, zolmitriptan, frovatriptan, sumatriptan.
  Other Names: Zomig® is a registered trademark of AstraZeneca; Maxalt® is a registered trademark of Merck & Co; Inc; Relpax® is a registered trademark of Pfizer; Frova® is a registered trademark of Elan Pharmaceuticals/UCB Pharma; Amerge® is a registered trademark of GlaxoSmithKline; Axert® is a registered trademark of Pharmacia; Imitrex® is a registered trademark of GlaxoSmithKline

SUMMARY:
The goal of this study is to measure medical resource utilization, treatment patterns, and costs for 1.) triptan-naïve patients with new pharmacy claims for a combination treatment of sumatriptan and naproxen sodium (SumaRT/Nap) or single-entity triptan and 2.) patients who are switched from one triptan to either SumaRT/Nap or a different single-entity triptan. The analysis will compare the mean number of prescription tablets used (including triptans, NSAIDs, opioids, and ergots) and migraine-specific medical resource utilization/costs and pharmacy costs incurred by health plan members who switched to SumaRT/Nap from a single-entity triptan. The null hypothesis for the triptan-naïve analysis is that no difference will be observed between resource utilization and costs incurred by patients treated with SumaRT/Nap and those treated with a single-entity triptan. The test hypothesis is that one group will incur significantly fewer costs and/or significantly lower health care utilization. For the triptan switch analysis, the null hypothesis is that no difference will be observed in the costs or health care utilization between triptan patients who are switched to SumaRT/Nap compared with those switched to a new triptan. The test hypothesis is that one treatment group will experience significantly lower costs and/or lower health care utilization.

The source of data for this analysis is the Lifelink Health Plan Claims Database (owned by IMS Health, Inc). This claims database includes more than 60 million covered lives. In addition to inpatient and outpatient records, this database includes standard and mail-order pharmacy claims with paid and charged amounts and dates of service.

Data from July 1, 2008 to December 31, 2009 (study period) will be used to conduct these retrospective analyses. Patients with at least one pharmacy claim for SumaRT/Nap between January 1, 2009 and June 30, 2009 (enrollment period) will be identified. The date of the first SumaRT/Nap pharmacy claim will be the index date for those patients. Each patient will be propensity score matched with an oral triptan patient based on the following pre-index covariates: age; gender; payer; geographic region; average monthly number of tablets of triptans, NSAIDs, and opioids; and average number of hospitalizations, emergency department visits, and physician visits in the month immediately preceding the index date as well as the mean number of hospitalizations, emergency department visits, and physician visits in the 5-month pre-index period. SumaRT/Nap patients and their single-entity matched controls who had no pharmacy claims for triptans prior to the index date will be analyzed in the triptan naïve group, and the SumaRT/Nap patients and their single-entity matched controls who switched to a new triptan will be analyzed in the switch analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 64 years
* Patients with continuous health plan eligibility during the 6-month pre-index period and follow-up period
* Patients in the triptan switch analysis must have at least one pharmacy claim for an oral triptan in the 6 month, pre-index period

Exclusion Criteria:

* Patients with a pharmacy claim for a nasal triptan at any time during the study period
* Patients with pharmacy claims for more than one type of oral triptan on the index date
* Patients in the single-entity oral triptan study groups who have a pharmacy claim for SumaRT/Nap during the 6-month follow-up period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be conducted using retrospective health care claims data from insured migraine patients aged 18 to 64. Patients with a pharmacy claim for a combination treatment of sumatriptan and naproxen sodium (SumaRT/Nap) during the index period will be identified. If the SumaRT/Nap prescription is not preceeded by a single-entity triptan pharmacy claim in the 6-month, pre-index period, that patient will be included in the triptan-naive cohort. Propensity score matching will be used to identify migraine patients with new single-entity triptan claims as a comparator group. Patients with a pharmacy claim for a single-entity triptan in the 6-month, pre-index period and a pharmacy claim for SumaRT/Nap will be included in the triptan switch cohort. Propensity score matching will be used to identify patients with similar characteristics who switch to a new triptan as a comparator group.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mean number of tablets dispensed | In the 6 months immediately preceding the index date and during the 6-month follow-up period that begins at the index date
  The mean number of tables dispensed as measured by pharmacy claims for prescription medications including triptans, NSAIDs, and opioids

SECONDARY OUTCOMES:
Mean and total migraine-related pharmacy costs | During the 6-month follow-up period that begins at the index date
  All costs will be adjusted to 2009 US dollars. Results will include costs to the health plan and costs to the patients. Costs will be reported for triptans, migraine prophylaxis, NSAIDs, opioids, and antiemetics
Mean and total migraine-related medical costs | During the 6-month follow-up period that begins at the index date
  All costs will be adjusted to 2009 US dollars. Costs will include those for hospitizations, emergency department visits, physician visits, other outpatient visits, and other medical costs
Mean numbers of migraine-related medical visits | During the 6-month follow-up period that begins at the index date
  Results will include hospitalizations, visits to the emergency department, physician visits, and other outpatient visits
Mean numbers and costs (adjusted to 2009 US dollars) of all-cause resource use measures | During the 6-month follow-up period that begins at the index date
  Results will include all-cause hospitalizations, emergency department visits, physician visits, and outpatient visits. Costs reported by total, pharmacy and medical
Presence of preventive medications | During the 6-month follow-up period that begins at the index date
  Pharmacy claims for migraine prophylactic medications including tricyclic antidepressants, calcium channel blockers, beta blockers, mirtazapine, venlafaxine, valproic acid, gabapentin, tiagabine, topiramate, carbamazapine, and botulinium toxin

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline